CLINICAL TRIAL: NCT00240760
Title: Efficacy and Safety of Memantine Hydrochloride, a Low Affinity Antagonist to N-Methyl-D-Aspartate (NMDA) Type Receptors, in the Prevention of Cognitive Decline and Disease Progression in Down's Syndrome
Brief Title: Memantine and Down's Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KCL/DS/MEM/1; EUDRACT- 2005 000381 39; ISRCTN47562898
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2006-02-20 (Estimated); Status verified 2005-10

CONDITIONS: Down's Syndrome; Dementia; Learning Disabilities
Keywords: Memantine; Down syndrome; Dementia; learning Disability; Treatment of Dementia
MeSH Terms: conditions — Down Syndrome; Dementia; Learning Disabilities | interventions — Memantine

INTERVENTIONS:
Drug: Memantine Hydrochloride

SUMMARY:
This is a study to assess whether memantine is effective and safe in preventing age related cognitive deterioration and dementia in people with Down's syndrome (DS) age 40 and over. The study will last for a year and it will include 180 people with Down's syndrome with and without dementia. Participants will be assessed on memory skills, attention and problem solving abilities. Quality of life and abilities for everyday living skills will also be regularly checked.

Primary Aims

Clinical:

* To determine the clinical efficacy of memantine versus placebo in preventing cognitive decline in people with DS.
* To compare the safety and tolerability of memantine versus placebo in people with Down's syndrome (DS).

Biochemical and pathological:

* To examine the ability of memantine to alter markers of disease progression in DS patients.

Secondary Aims

Clinical:

* To determine whether memantine has, as compared with placebo, a significant positive impact on:

  * level of independent functioning as measured by the carer-rated adaptive behavioural scale, (ABS) in adults with DS;
  * quality of life in adults with DS.

Biochemical and pathological:

* To investigate putative markers of memantine's mechanism of action in peripheral samples from living patients with DS.

DETAILED DESCRIPTION:
Over the age of 40, all people with Down's Syndrome have substantial changes in the brain similar to those of Alzheimer's disease and most are at very high risk of developing a clinical dementia with progressive decline of function and cognitive abilities.

There are changes to all of the key chemical messenger systems in the brain as people develop Alzheimer's disease. One of the most ubiquitous chemical messenger systems, present on the majority of nerve cells in the brain, is called the glutamatergic system. In this system the main receptors present on the nerve endings are referred to as glutamate receptors. Under certain circumstances, usually when there is damage to particular parts of the brain, these receptors can lead to "overfiring" of the nerve cells with disastrous consequences. This can result in the generation of a number of toxic chemical molecules that lead to further damage to the nerve cells (such as phopholipases, proteases, nitric oxide synthases, inflammatory molecules and free radicals), usually referred to as excitotoxicity. Memantine blocks the effects of pathologically elevated tonic levels of glutamate that may lead to dysfunction of nerve cells and in this way is thought to block the main glutamate excitotoxicity site on nerve cells.

Randomized clinical trials in people with Alzheimer's disease indicate that memantine significantly slows down the progression of functional and cognitive impairments. Memantine has now been licensed for the treatment of moderate-severe Alzheimer's disease on the basis of these trials. We would hypothesise that older people with Down's syndrome would particularly benefit from treatment with Memantine, partly because of the large amount of Alzheimer's disease changes present in the brain and partly because excessive glutamate receptor activity has been demonstrated in adults with Down's syndrome.

In a recent study we assessed 122 individuals with Down's Syndrome using newly developed neuropsychometric battery of tests, (the the Down's syndrome Attention, Memory and Executive function battery -DAME battery, Margallo-Lana 2002a,b). People with Down's Syndrome over the age of 40 without dementia experienced a decline of 11% over one year, indicating that progressive cognitive decline precedes dementia (hence offering an important opportunity for prevention) and that these measurements are sensitive to cognitive change over time, hence a trial to evaluate the prevention of dementia is feasible with current evaluation measures.

Study Design:

Participants will be given Memantine or placebo (dummy tablet) for 52 weeks. To avoid bias, participants will be allocated to the placebo or Memantine group at random (this is a randomized trial) and none of the researchers or participants will know which treatment people are getting (the study is double blind). However, in an emergency, the investigators can contact the study pharmacist to find out whether a particular participant was receiving Memantine or the dummy tablet. The placebo and Memantine groups will be compared at the end of the study (the study is placebo control) to see if Memantine is any better than the dummy pill. The efficacy of Memantine will be assessed by comparing the change in scores between the initial assessments and assessments in the follow-up period at 12, 26 and 52 weeks. Thus participant will be assessed on 4 occasions.

Assessments:

In addition to a clinical history and the collection of standardized information such as any adverse events, the assessment will include:

1. Assessment of memory, attention and planning abilities:

   Memory, attention and executive function (planning abilities) will be assessed by direct testing with the participants using the DAME battery. The DAME battery has been validated as a measure that is sensitive to change in older people with Down's syndrome. The range of scores is 0-241 and can be completed in 45 minutes by most people with mild-moderate learning disability. The test re-test and inter-rater reliability is XX and YY respectively.
2. Development of dementia:

   To facilitate the diagnosis of dementia, we will use the Dementia Questionnaire for mentally Retarded Persons (DMR). This is a standardised, validated and reliable tool specifically developed to aid the assessment of dementia in people with mild and moderate learning disabilities. It is an informant-based questionnaire and consists of 50 items to be completed by family or staff about the patient who is known to them. Items are arranged in 8 subscales: short term memory; long-term memory; spatial and temporal orientation; speech; practical skills; mood; activity and interest; behaviour and disturbance. The range of scores is 0-104 and can be completed in 15-20 minutes. The inter-rater reliability is 0.76.
3. Diagnosis of dementia:

   Standardized criteria for diagnosis of dementia based on the International Classification of Diseases, 10th Version (ICD 10) will be used by 2 experts (Dr Margallo-Lana, Dr Prasher) to identify new cases. The assessment for dementia will be done at baseline, week 26 and week 52 assessments.

   The diagnosis of dementia will be based on clinical information supplied by carers aided by the use of the Dementia Questionnaire for Persons with Mental Retardation (DMR).
4. Independent functioning :

   Independent functioning will be evaluated using the Adaptive Behavioural Scale (ABS, Nihira,1974). This is an informant based instrument and is part of the assessment used by the American Association on Mental Deficiency (Nihira, 1974) to assess daily living skills in people with learning disabilities. The ABS measures ten groups of skills related to self-care and socialization. The ten skills groups: independent functioning, physical development, economic activity, language development, numbers and time, domestic activity, vocational activity, self-direction, responsibility, and socialization. The ABS has a test-retest reliability of .96, which is very good. Score range is 0-280.
5. Quality of life:

   Quality of life will be evaluated with the Quality of Life in Alzheimer's Disease (Logsdon et al. 1998). This scale was specifically developed to measure quality of life in people with dementia. It is composed of 13-items that measure physical condition, mood, memory, functional abilities, interpersonal relationships, ability to participate in meaningful activities, financial situation, and global assessments of self as a whole and QOL as a whole. The response options are 4-point multiple choice options (1 = poor, 4 = excellent). Scale scores range from 13 to 52, with higher scores indicating greater QOL.
6. Global change:

   The Clinician's Global Impression of Change (CGI/C) has been one of the most commonly used test to assess overall change in clinical trials (Guy, 1976). The validity of this type of measure is based on the ability of an experienced clinician to detect clinically relevant against trivial change in a patient's overall clinical state. These simple scales have been shown to be remarkably sensitive to change in cholinesterase inhibitor trials (Schneider, 1997).
7. Standardized schedule to monitor any side effects/adverse events.

Participants:

180 people aged > 40 with DS (with or without dementia) who have mild-moderate learning disability, in a double blind, placebo controlled design.

Related Biochemical Studies:

Blood samples (10ml) will be taken at baseline and the final follow-up assessment. Blood will be processed to yield four different components: plasma, platelets, red and white blood cells.

Plasma concentrations of the amino acid neurotransmitters aspartate and glutamate will be measured together with the rate of uptake of glutamate into blood cells (platelets). The ability of glutamate to bind to the platelets' receptors (particularly the NMDA receptor - a sub-type of glutamate receptor) will also be also assessed. These investigations will determine whether Memantine protects and modulates glutamatergic transmission.

Plasma concentrations amyloid (Abeta species 1-40/1-42), the protein that typically accumulates in the brains of people with Alzheimer's disease, will also be measured together with plasma concentrations of the amyloid precursor protein (APP). Preliminary studies will be also undertaken to see if glutamate receptors in platelets (NMDA receptors) regulate the release of APP/Abeta.

The study will also investigate genetic factors that may affect the risk of Alzheimer's disease in people with Down's Syndrome. Any identified genetic factors will be examined to see if they can predict response to treatment.

These investigations will help to determine if Memantine alters the accumulation of proteins in the brain typical of Alzheimer's disease in people with Down's syndrome.

Consumers panels of relatives of people with DS and carers have been involved in protocol development and the writing of information sheets.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be:

1. Participants with learning disabilities due to Down's syndrome (DS) confirmed by karyotype. A clinical diagnosis (provided by the participant's general practitioner or hospital specialist) will be accepted if karyotype is not known and participant does not agree to have it tested
2. Ages 40 years and over or any age if a diagnosis of dementia is established
3. In participants with dementia, the diagnosis will be consistent with the 10th version of the International Classification of Diseases (ICD-10) (World Health Organization [WHO], 1992) diagnostic criteria
4. Level of speech and comprehension of verbal commands are sufficient to understand and to answer simple requests
5. Resident in care facility or community living with a carer who is willing to accept responsibility for supervising the treatment and will provide input to efficacy parameters in accordance with protocol requirements
6. Not receiving treatment with memantine currently or in past 4 weeks and responsible clinician not considering treatment with memantine
7. Participant willing to take part in study; and carer, with capacity, willing to assent to study and agrees that participant can take part if participant is also willing.

Exclusion Criteria:

Exclusion criteria will be:

1. Participants known to have sensitivity to memantine
2. Severe, unstable or uncontrolled medical or psychiatric conditions apparent from history, physical examination or investigations
3. A current diagnosis of primary neurodegenerative disorder other than dementia such as Huntington's disease, etc.
4. Uncontrolled epilepsy
5. Presence of challenging behaviour likely to preclude the participation during testing
6. Presence of severe motor or sensory impairment (severe deafness or blindness) that renders the participant as untestable with the battery of tests used in the study
7. Current evidence of delirium
8. Severe renal impairment
9. Low probability of treatment compliance
10. Previous evidence of lack of efficacy or tolerability to memantine
11. Taking any of the following substances:

    * an investigational drug during the 4 weeks prior to randomization
    * a drug known to cause major organ system toxicity during the 4 weeks prior to randomization
    * started any new psychotropic during the 4 weeks prior to randomization; participants who had been on a stable dose of psychotropic during the 4 weeks prior to randomization are still eligible.
    * memantine during the 6 weeks prior to randomization
    * other N-methyl-D-aspartate (NMDA) antagonists: amantadine, ketamine, and dextromethorphan
    * barbiturates and primidone
    * baclofen and dantrolen
    * dextromethorphan
    * antimuscarinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2005-10

PRIMARY OUTCOMES:
Down's Attention Memory and Executive Function Scale
Part I of the Adaptive Behaviour Scale

SECONDARY OUTCOMES:
The Quality of Life in Alzheimer's Disease (Logsdon et al. 1998)
Clinician's Global Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Verinder Prasher, PhD, Principal Investigator — King's College London; Clive G Ballard, Professor, Study Director — King's College London; Paul Francis, PhD, Principal Investigator — King's College London; Ed Juszczak, PhD, Principal Investigator — University of Oxford; Jill Mollis, PhD, Principal Investigator — University of Oxford; Maria Luisa Margallo-Lana, PhD, Principal Investigator — Northgate and Prudhoe NHS Trust
Locations (2):
- United Kingdom (2):
  - Monyhull Hall Road, Birmingham, Birmingham
  - Northgate Hospital, Morpeth, Northumberland